CLINICAL TRIAL: NCT03540277
Title: The Effect of Addition of Parental Component to the Program "Young In Favor of Myself" on Participating Parents and Their Children
Brief Title: Prevention Program- Promoting Self Resilience, Positive Self-Image and Body Image Among Adolescents and Their Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Hai College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Tel Hai College.
Record Dates: First submitted 2018-04-26; First posted 2018-05-30 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Primary Prevention
Keywords: prevention program; body-image; self-esteem; parents; adolescents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prevention Program "young In Favor of Myself", active parents (Experimental): The program "young In Favor of Myself" will be delivered to adolescence aged 10-12, over 3 months. The program contains nine weekly, 90-min sessions that focus on Media literacy, self-esteem, self-image and body image. The parents will also participate by a phone app that will pass the parents activities to do with their children, in parallel to the program. All participants will complete a self-report questionnaire at baseline, after the program ends, and three months after the completion of the program.
  Interventions: Behavioral: Experimental: Prevention Program "young In Favor of Myself", active parents
- Prevention Program "young In Favor of Myself", passive parents (Active Comparator): The program "young In Favor of Myself" will be delivered to adolescence aged 10-12, over 3 months. The program contains nine weekly, 90-min sessions that focus on Media literacy, self-esteem, self-image and body image. The parents won't participate in the program, they will get only a brochure about Media literacy, self-esteem, self-image and body image. All participants will complete a self-report questionnaire at baseline, after the program ends, and three months after the completion of the program.
  Interventions: Behavioral: Experimental: Prevention Program "young In Favor of Myself", no parental involvement
- control group (No Intervention): The control group will not receive the intervention program. The control group will complete the same self-report questionnaire as the intervention group at baseline, after the program ends, and three months after the completion of the program.

INTERVENTIONS:
Behavioral: Experimental: Prevention Program "young In Favor of Myself", active parents — Prevention program: "young In Favor of Myself", with parent participation
  Arms: Prevention Program "young In Favor of Myself", active parents
Behavioral: Experimental: Prevention Program "young In Favor of Myself", no parental involvement — Prevention program: "young In Favor of Myself", without parent participation
  Arms: Prevention Program "young In Favor of Myself", passive parents

SUMMARY:
Cluster-Randomized Clinical trial, which includes the development and activation of an intervention program among young adolescents and their parents. Study hypothesis is that the intervention program will yield improvement in adolescents whose parents participated in the program, in comparison with the adolescents whose parents weren't involved in the intervention. Results will be measured using the study questionnaire, to be filled out by the participants before, after, and three months after the completion of the program. The questionnaire will include validated questionnaires with good psychometric qualities. The study protocol was approved by Tel Hai College institutional review board. Parents of all participants, in the intervention and in the control group, received information about the program and the study and were asked to provide informed consent.

DETAILED DESCRIPTION:
Early adolescent (10-13 years) is characterized by hormonal changes and accelerated physiological growth. Significant risk factors for the physical and mental health of children and adolescents include, among other things, disordered eating patterns, overweight and reduced physical activity, low self-esteem and negative body image.

"In Favor of Myself" is a preventive intervention program. The program's primary goal is to increase adolescents' self-esteem and to prevent negative self-image and body image, as well as to development media literacy. In this study, the investigators will focus on the "Young In Favor of Myself " program, designed for ages 10-12, grades 5 and 6, and its main core is the development of self-care. To increase the effect of "Young In Favor of Myself " program, on the adolescents, the investigators have developed a program that will be passed on to parents through a telephone application. The study will first assess the parents' influence on the program, and then evaluate the difference in adolescent outcomes from the program with or without this supplement.

Results will be measured using the study questionnaire, to be filled out by the participants (both parents and adolescents) before, after, and three months after the completion of the program. The questionnaire will include validated questionnaires with good psychometric qualities. The study protocol was approved by Tel Hai College institutional review board. Parents of all participants, in the intervention and in the control group, received information about the program and the study and were asked to provide informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children 10-12 years old
* 10-12-year-old children of participating parents
* Participants who filled out the questionnaires before and after the program
* Participants whose parents signed a letter of informed consent.

Exclusion Criteria:

• Participants who didn't complete the questionnaires at baseline or at least twice.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Sociocultural Attitudes towards Appearance Questionnaire-4, Affects by Media subscale. | Measured three times over six months: at baseline, after the program ends, and three months after the completion of the program, measuring a change in scores
  The Sociocultural Attitudes Towards Appearance Questionnaire (Schaefer et al., 2015). The investigators included the Media subscale, including 4 items. Items are rated on a 5-point scale: (1) always, (2) often, (3) sometimes, (4) rarely, (5) never. The total score is based on computing the average. A higher score indicates higher pressure from the media to change one's look.
Change from Baseline in Rosenberg Self Esteem Scale | Measured three times over six months: at baseline, after the program ends, and three months after the completion of the program, measuring a change in scores
  Rosenberg Self Esteem Scale (Rosenberg, 1965)- 10 items. Scoring involves a method of combined ratings. Low self-esteem responses are "disagree" or "strongly disagree" on items 1, 3, 4, 7, 10, and "strongly agree" or "agree" on items 2, 5, 6, 8, 9. Two or three out of three correct responses to items 3, 7, and 9 are scored as one item. One or two out of two correct responses for items 4 and 5 are considered as a single item; items 1,8, and 10 are scored as individual items; and combined correct responses (one or two out of two) to items 2 and 6 are considered to be a single item.
Change from Baseline in Body Esteem Scale | Measured three times over six months: at baseline, after the program ends, and three months after the completion of the program, measuring a change in scores
  Body Esteem Scale- This questionnaire examines self-esteem of body and physical appearance and consists of 3 subscales: appearance (10 items), weight (8 items) and attribution 187 to others (5 items). Items are rated on a 5-point scale: (1) never, (2) rarely, (3) sometimes, (4) 188 often, and (5) always. A higher score indicates higher body-esteem (Mendelson, Mendelson, & White, 2001)
Change from Baseline in Eating Disorder Examination- Questionnaire (EDE-Q8) | Measured three times over six months: at baseline, after the program ends, and three months after the completion of the program, measuring a change in scores
  Eating Disorder Examination- Questionnaire short version (EDE-Q8). The items are rated on a 6-point scale: (1) never, (2) rarely, (3) sometimes, (4) often, (5) usually, and (6) always. EDE-Q provides assessment of eating disorder psychopathology related to anorexia nervosa (AN), bulimia nervosa (BN), and binge-eating disorder (BED). (Kliem et al, 2016)
Change from Baseline in Advertising Scale | Measured three times over six months: at baseline, after the program ends, and three months after the completion of the program, measuring a change in scores
  The Advertising scale contains 1 item- Identification of strategies used by media. This question is reflected as a protective factor. It contains 8 different strategies which participants choose from: higher number of strategies identified indicate better media literacy. (Golan et al., 2013).
Change from Baseline in Self-Caring | Measured three times over six months: at baseline, after the program ends, and three months after the completion of the program, measuring a change in scores
  Developed by Prof. Moria Golan and assessed in previous research. Includes 14 items which are rated on a 4-point scale: (1) never, (2) rarely, (3) sometimes, (4) always. Items are summed, and higher scores indicate higher self-care behaviors. This questionnaire was designed to assess self care behaviors in adolescents.

SECONDARY OUTCOMES:
The 11-item Knowledge Test BEC | Measured three times over six months: at baseline, after the program ends, and three months after the completion of the program, measuring a change in scores
  The 11-item Knowledge Test BEC was developed to assess knowledge of parenting strategies to prevent unhealthy eating and body dissatisfaction in young children. Scores are summed across the 11 items giving a total score ranging between 11 and 44, with higher scores indicating greater knowledge of parenting strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Moria Golan, Prof., Principal Investigator — Tel Hai College
Locations (1):
- Tel Hai Academic College, Kiryat Shmona, North of Israel, Israel

REFERENCES:
- [Derived] Golan M, Benifla S, Samo A, Alon N, Mozeikov M. Feasibility and effect of adding a concurrent parental component to a school-based wellness program using two modes of mobile-based technology - mixed methods evaluation of RCT. BMC Public Health. 2022 Feb 14;22(1):297. doi: 10.1186/s12889-022-12581-7. PMID 35164721